CLINICAL TRIAL: NCT03149419
Title: Endothelial, Autonomic and Pressure Effects of Paroxetine in Recent Postmenopause Women With Hot Flashes: a Randomized Placebo Controlled Clinical Trial
Brief Title: Hot Flash as a Marker of Cardiovascular Risk in Recent Postmenopause: Effects of Non-hormonal Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Ciciliana Maíla Zilio Rech, Principal Investigator, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 6717515.1.0000.5259
Record Dates: First submitted 2017-04-18; First posted 2017-05-11 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Postmenopausal Flushing; Cardiovascular Risk Factor; Endothelial Dysfunction
Keywords: postmenopause; paroxetine; endothelial dysfunction; blood pressure; heart rate variability; sleep quality; perceived stress; sleepiness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleepiness | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paroxetine (Active Comparator): Paroxetine 7,5 mg - 1 pill/day for 12 weeks
  Interventions: Drug: Paroxetine
- Placebo (Placebo Comparator): Placebo oral capsule (corn starch) - 1 pill/day for 12 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Paroxetine
  Arms: Paroxetine
Drug: Placebo oral capsule
  Arms: Placebo

SUMMARY:
Hot flashes, vasomotor symptoms that affect many postmenopausal women, are associated with cardiovascular disease and endothelial dysfunction. Estrogen therapy, associated or not with progestogens, is the standard treatment for vasomotor symptoms and improves the endothelial function of postmenopausal women with hot flushes, even those with cardiovascular risk factors, such as hypertension. It is not known whether hot flushes are a cause for the development of endothelial dysfunction or are markers of this dysfunction, evidenced by estrogen deficiency, thus representing primitive target organ (vessel) lesion. Paroxetine was approved by the FDA as a non hormonal treatment for menopausal hot flashes. In this double-blind randomized clinical trial, the vascular effects of paroxetine at a dose of 7.5 mg / day, compared to placebo, during 12 weeks are evaluated.

DETAILED DESCRIPTION:
Paroxetine and placebo effects at baseline and after 12 weeks in endothelial, autonomic and pressure components of vascular function are evaluated.

Non invasive venous occlusion plethysmography is used to study endothelial function; ambulatory blood pressure monitoring is used to study blood pressure variations during daytime and nocturnal descent; autonomic function is studied following sympathetic and parasympathetic parameters through heart rate variability.

The effects of paroxetine and placebo are also evaluated on:

* daytime sleepiness (through Epworth Sleepiness Scale ),
* sleep quality (through Pittsburgh Sleep Quality Index),
* perceived stress (through Perceived Scale Stress).

Biochemical and hormonal profiles including complete lipid profile, fasting glucose, insulin, estradiol, follicle stimulating hormone (FSH), luteinizing hormone (LH); inflammatory and oxidative stress markers are also studied.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopause
2. Present hot flushes (note ≥ 3 on a scale of 0 to 10)

Exclusion Criteria:

1. > 10 years of hypoestrogenism
2. Smoking
3. Diabetes mellitus or altered fasting glycemia in use of oral hypoglycemic agents or insulin
4. BMI ≥ 35 Kg / m2
5. Uncontrolled hypertension - blood pressure (BP) ≥ 140/90 mmHg
6. Users of glucocorticoids, phytoestrogens, β-blockers, selective serotonin reuptake inhibitors (SSRIs), selective noradrenaline reuptake inhibitors (SNRIs), clonidine, gabapentin, pregabalin, cinnarizine, alphamethyldopa or any drugs with effects on the central nervous system;
7. Uncompensated hypo or hyperthyroidism;
8. Previous cardiovascular event history.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Endothelial function in non invasive venous occlusion plethysmography | 12 weeks
  Forearm blood flow (ml/min per 100 ml)

CONTACTS AND LOCATIONS:
Overall Officials: Ciciliana MZ Rech, Principal Investigator — Universidade do Estado do Rio de Janeiro- BioVasc laboratory; Ruth Clapauch, PhD, Study Chair — Rio de Janeiro State University
Locations (1):
- Universidade do Estado do Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taddei S, Virdis A, Ghiadoni L, Mattei P, Sudano I, Bernini G, Pinto S, Salvetti A. Menopause is associated with endothelial dysfunction in women. Hypertension. 1996 Oct;28(4):576-82. doi: 10.1161/01.hyp.28.4.576. PMID 8843881
- [Background] Bechlioulis A, Kalantaridou SN, Naka KK, Chatzikyriakidou A, Calis KA, Makrigiannakis A, Papanikolaou O, Kaponis A, Katsouras C, Georgiou I, Chrousos GP, Michalis LK. Endothelial function, but not carotid intima-media thickness, is affected early in menopause and is associated with severity of hot flushes. J Clin Endocrinol Metab. 2010 Mar;95(3):1199-206. doi: 10.1210/jc.2009-2262. Epub 2010 Jan 15. PMID 20080857
- [Background] Lambrinoudaki I, Augoulea A, Armeni E, Rizos D, Alexandrou A, Creatsa M, Kazani M, Georgiopoulos G, Livada A, Exarchakou A, Stamatelopoulos K. Menopausal symptoms are associated with subclinical atherosclerosis in healthy recently postmenopausal women. Climacteric. 2012 Aug;15(4):350-7. doi: 10.3109/13697137.2011.618564. Epub 2011 Dec 1. PMID 22132748
- [Background] Silveira JS, Clapauch R, Souza Md, Bouskela E. Hot flashes: emerging cardiovascular risk factors in recent and late postmenopause and their association with higher blood pressure. Menopause. 2016 Aug;23(8):846-55. doi: 10.1097/GME.0000000000000641. PMID 27219834
- [Background] Orleans RJ, Li L, Kim MJ, Guo J, Sobhan M, Soule L, Joffe HV. FDA approval of paroxetine for menopausal hot flushes. N Engl J Med. 2014 May 8;370(19):1777-9. doi: 10.1056/NEJMp1402080. No abstract available. PMID 24806158